CLINICAL TRIAL: NCT01063842
Title: Tolerability Improvement of Tramadol/Acetaminophen (Ultracet) by Titration in Korean OA Patients:Multicenter, Randomized, Double-blind Study
Brief Title: A Study of the Tolerability of Titrated Dose Tramadol/Acetaminophen Combination Tablet in Korean Patients With Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Medical Director, Janssen Korea, Ltd., Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004990
Record Dates: First submitted 2009-10-08; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Osteoarthritis
Keywords: Drop-out rate; Osteoarthritis; Tolerability; Tramadol; Acetaminophen
MeSH Terms: conditions — Osteoarthritis | interventions — Ultracet; Tramadol; Acetaminophen

ARMS (2):
- 001 (Experimental): tramadol hydrochloride / acetaminophen and placebo 1 tablet of tramadol/acetaminophen in the morning 1 tablet of placebo in the afternoon and evening for 3 days then 1 tablet of tramadol/acetaminophen in the morning evening and 1 tablet of placebo in the afternoon for 4 days then 1 tablet of tramadol/acetaminophen 3 times daily for next 7 days
  Interventions: Drug: tramadol hydrochloride / acetaminophen and placebo
- 002 (Active Comparator): tramadol hydrochloride /acetaminophen 1 tablet of tramadol hydrochloride/acetaminophen three times daily without titration for 14 days.
  Interventions: Drug: tramadol hydrochloride /acetaminophen

INTERVENTIONS:
Drug: tramadol hydrochloride /acetaminophen — 1 tablet of tramadol hydrochloride/acetaminophen three times daily without titration for 14 days.
  Arms: 002
Drug: tramadol hydrochloride / acetaminophen and placebo — 1 tablet of tramadol/acetaminophen in the morning, 1 tablet of placebo in the afternoon and evening for 3 days, then 1 tablet of tramadol/acetaminophen in the morning, evening and 1 tablet of placebo in the afternoon for 4 days, then 1 tablet of tramadol/acetaminophen 3 times daily for next 7 days
  Arms: 001

SUMMARY:
The purpose of this study is to compare the number of osteoarthritis patients receiving titrated or increasing doses of tramadol hydrochloride/acetaminophen combination tablet (titration group) who discontinue treatment due to adverse events to the number of patients receiving a non-titrated dose of tramadol/hydrochloride/acetaminophen combination tablet who discontinue treatment due to adverse events.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), multicenter, double-blind (neither physician nor patient knows the name of the assigned drug), add-on study (NSAIDs or COX-2 medications maintained at pre-study dose.) to investigate the tolerability of titrated doses of tramadol hydrochloride/acetaminophen combination tablet in osteoarthritis patients taking NSAIDS or COX-2 inhibitors (both are drugs used to treat inflammation and pain) compared to non-titrated doses of tramadol hydrochloride/acetaminophen combination tablet. The patients will be randomized into 2 treatment groups. First group (the titration group) receives 1 tablet of tramadol hydrochloride/acetaminophen in the morning, 1 tablet of placebo in the afternoon and evening for 3 days, then 1 tablet of tramadol hydrochloride/acetaminophen in the morning, 1 tablet of placebo in the afternoon and 1 tablet of tramadol hydrochloride/acetaminophen in the evening for 4 days, and the 1 tablet of tramadol hydrochloride/acetaminophen three times daily for next 7 days. The second group (non-titration group) will receive 1 tablet of tramadol hydrochloride/acetaminophen three times daily without titration for 14 days. The study hypothesis is the first group's discontinuation rate due to adverse events is lower than that of second group. Safety assessments include adverse event, vital sign and clinical lab monitoring. First group will receive 1 tablet of tramadol hydrochloride/acetaminophen and 2 tablets of placebo for 3 days, 2 tablets of tramadol hydrochloride/acetaminophen and 1 tablet of placebo for 4 days, and 3 tablets of tramadol hydrochloride/acetaminophen for 7 days. Second group will receive 3 tablets of tramadol hydrochloride/acetaminophen for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have osteoarthritis of the knee for at least one year based on clinical and radiological criteria
* Must have been on a stable daily dose of a NSAID for at least two weeks prior to randomization
* Must have a pain intensity Numeric Rating Scale (NRS) score 4 or more as a average intensity for 48 hours. (On a Numeric Rating Scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable)

Exclusion Criteria:

* Have taken tramadol HCL within 14 days prior to randomization
* Have taken acetaminophen within 7 days prior to randomization
* Have received other pain medication (including topical medication and/or anesthetics), sedative hypnotics, or muscle relaxants within a period of less than five half-lives of the given medication prior to randomization

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-08; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Study Discontinuation rate due to adverse event | Throughout the study from start of study drug until final visit, Day 14

SECONDARY OUTCOMES:
comparison of the pain intensity scores between the 2 treatment groups | Day 0, Day 14
comparison of the pain relief scores between the 2 treatment groups | Day 14
comparison of the WOMAC (Western and Ontario Mcmaster) total scores between the 2 treatment groups.The WOMAC index is a 24-item questionnaire completed by the patient and focusing on pain, stiffness and function related to osteoarthritis of knee and hip | Day 0, Day 14
comparison of the overall assessment of patient between the 2 treatment groups | Day 14
comparison of the overall assessment of investigator between the 2 treatment groups | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.